CLINICAL TRIAL: NCT02154308
Title: A Multicenter, Open-Label, Phase 3 Clinical Study to Evaluate the Immunogenicity and Safety of IL-YANG Inactivated Split Influenza Vaccine in Healthy Adults 18 to < 65 Years of Age and in Healthy Adults ≥ 65 Years of Age.
Brief Title: Phase 3 Study to Evaluate the Immunogenicity and Safety of Inactivated Split Influenza Vaccine in Healthy Korea Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IY_IFEZ_AD_301
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Influenza; Influenza vaccine; Split influenza vaccine; Seasonal influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IL-YANG influenza vaccine (Experimental): IL-YANG FLU Vaccine Prefilled Syringe INJ 0.5mL by intramuscular injection
  Interventions: Biological: IL-YANG FLU Vaccine Prefilled Syringe INJ 0.5mL

INTERVENTIONS:
Biological: IL-YANG FLU Vaccine Prefilled Syringe INJ 0.5mL — IL-YANG FLU Vaccine Prefilled Syringe INJ 0.5mL by intramuscular injection

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of IL-YANG Inactivated Split Influenza Vaccine (IL-YANG FLU Vaccine Prefilled Syringe INJ.) administered as a single intramuscular injection.

DETAILED DESCRIPTION:
This is a multicenter, open-label study. Subjects who have provided written informed consent will undergo the protocol-specific assessments to determine their eligibility for the study. Subjects considered eligible will be assigned to an appropriate age stratum, and will be given a single dose of the study vaccine. For each age stratum, the first 142 subjects enrolled will be evaluated for both immunogenicity and safety, and the remaining subjects subsequently enrolled will be evaluated only for the safety of the study vaccine.

1. Group A: healthy adults 18 to < 65 years of age
2. Group B: healthy adults ≥ 65 years of age

The investigator will evaluate the immunogenicity and safety of the study vaccine throughout the study. The immunogenicity assessment will be performed at Visit 1 (pre-vaccination) and at the End-of-Study Visit. For safety measurements, subjects will be instructed to record any adverse events occurring after vaccination in the Patient Diary card.

Subjects who are assigned for the both immunogenicity and safety assessment will have their blood sample drawn for antibody titer (immunogenicity) testing, and afterward, receive 0.5 mL of the study vaccine by intramuscular injection at deltoid muscle. Subjects will return to the clinic for follow-up visit 4 to 5 weeks after the vaccination, and undergo another blood sampling for antibody titer test. The long-term safety for up to 6 months after vaccination will be also evaluated. Subjects who are assigned for only safety assessments will not undergo blood sampling, but have the same visit schedule as those assigned for the both immunogenicity and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man and woman 18 years of age or older
* Woman of childbearing potential must have a negative urine human chorionic gonadotropin (HCG) test at screening
* Subject who was given, and fully understood, the information about the study, made a voluntary decision, and provided written informed consent, to participate in the study and comply with all applicable study requirements.

Exclusion Criteria:

* Subject with a known allergy to eggs, chicken, neomycin, gentamicin or any components of the study vaccine
* Subject who had received an influenza vaccine within the last 6 months
* Subject who has, or has a family history of, an immune system disorder including immune deficiency disease
* Subject who had participated in blood donation within 1 week prior to vaccination, or is planning to participate in blood donation from Day 1 until Month 7 post-vaccination.
* Subject with a history of Guillain-Barre syndrome
* Subject with Down's syndrome or cytogenetic disorders.
* Subject with severe chronic disease which in the investigator's opinion would not make the subject a good candidate for the clinical trial
* Subject with hemophilia or being treated with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection
* Subject who had an acute fever with body temperature > 38.0 Cº within 72 hours prior to administration of the study vaccine
* Subject who had received any product containing acetylsalicylic acid or aspirin within 14 days prior to administration of the study vaccine
* Subject who had previously received another vaccine within 28 days before administration of the study drug, or is scheduled to receive another vaccine during the study period.
* Subject who had received immunosuppressant or immune modifying drug within the last 3 months prior to administration of the study vaccine
* Subject who had previously received immunoglobulin or blood-derived products within the last 3 months prior to administration of the study vaccine, or is expecting to be treated with immunoglobulin or blood-derived products during the study.
* Subject who had participated in another experimental study within 30 days prior to administration of the study vaccine
* Woman of childbearing potential at screening or woman who plans to become pregnant during the study. A woman of childbearing potential must have a negative pregnancy test, and, unless surgically sterile, must use an effective method of contraception throughout the study to be eligible for the study. Periodic abstinence and withdrawal are not considered as acceptable methods of contraception. Use of hormonal contraceptives is not allowed.
* Subject with other clinically significant medical or psychological condition who in the investigator's opinion would not be suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Solicited local & general Adverse Event, Unsolicited Adverse Event | up to Day28(+7)
  Solicited local reaction: pain, tenderness, redness, swelling Solicited general reactions: fever, nausea/vomiting, diarrhea, headache, fatigue, myalgia
Percentage of subjects achieving seroconversion and seroprotection for HI antibody after administration of the study vaccine | up to Day28(+7)
  Seroconversion: a pre-vaccination (Day 0) hemagglutination-inhibition (HI) antibody titer < 1:10 and a post-vaccination (Day 28) HI antibody titer ≥ 1: 40 (Case 1), or a pre-vaccination (Day 0) HI antibody titer ≥ 1:10 and a minimum four-fold rise in post-vaccination (Day 28) HI antibody titer (Case 2).
  Seroprotection: post-vaccination (Day 28) HI antibody titer ≥ 1:40

SECONDARY OUTCOMES:
Physical examination finding, vital signs | Day28(+7)
Geometric Mean Titer (GMT) of HI antibody titer before vaccination and after vaccination | Day28(+7)
  Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR), as measured by pre-vaccination (Day 0) HI antibody titer and post-vaccination (vaccination + 28 days) HI antibody titer.
Percentage of subjects with a pre-vaccination (Day 0) HI antibody titer < 1:40, and a minimum four-fold rise in post-vaccination (Day 28) HI antibody titer | Day28(+7)

CONTACTS AND LOCATIONS:
Overall Officials: IL-YANG PHARM, Study Director — IL-YANG Pharmaceutical Co.,LTD
Locations (1):
- Incheon St. Mary's Hospital, The Catholic University of Korea etc, Total 10 hospitals., Seoul Etc, South Korea